CLINICAL TRIAL: NCT00722657
Title: Social-Economics Profile of the Asthmatic Patients Attended at Nucleus of Integrated Medical Care
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Responsible Party: Social-economics Profile of the Asthmatic Patients attended at Nucleus of Integrated Medical Care, Fortaleza University
Other Study IDs: 08-004
Record Dates: First submitted 2008-07-22; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-05

CONDITIONS: Asthmatic Patients
Keywords: asthma; epidemiology
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: None Retained — None Retained - no samples retained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study had a descriptive, retrospective, transversal character with quantitative approach, which aimed to delineate the social-economics profile of the asthmatic patients that used the health service available at the Care Nucleon Medical Integrate (NAMI)

DETAILED DESCRIPTION:
The need of studies to develop programs of pharmaceutical attention for asthmatics was given because of the increase of incidence and prevalence of the disease in the population. This study had a descriptive, retrospective, transversal character with quantitative approach, which aimed to delineate the social-economics profile of the asthmatic patients that used the health service available at the Care Nucleon Medical Integrate (NAMI). The studied population was composed of 40 asthmatic patients who attended between April and May, during 2006. Data collection was performed through a semi-structured stereotypic questionnaire, with closed and opened questions. The age range of the interviewee between 0 to 5 years old represents the biggest percentage of patients, obtaining 60% of the answered questionnaires. According to social-economics conditions, 55% were illiterate or were learning to read, 75% were using some drug prescribed at NAMI, 72.5% deny completely the disease, 52.5% recognized the factors that triggered the asthmatic crisis and 55% said having often crisis. Seventy per cent (70%) of the interviewee showed some difficulty related to the use of the drugs; 47.5% have different problems related to the access to the medications. Through the analysis of the social-economics profile delineated of the asthmatics patients attended at NAMI, it could be revealed that the biggest part of the patients are people with little instruction, due to the social exclusion in which they are found; being the majority of them children of the female gender.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in regular Nucleus of Integrated Medical Care;
* Patients presented within the age group above to 80 years;
* Patients accepted voluntarily join the search;
* They used any medicine that received at the pharmacy of Nucleus of Integrated Medical Care.

Exclusion Criteria:

* Patients who don´t residing in the neighborhood of community;
* Patients who don´t accepted part of the study by answering the questionnaire;
* Have not made use of medicines in the last 60 days or have not received in the pharmacy of of Integrated Medical Care.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anísia T. Praxedes, yes, Principal Investigator — Fortaleza University